CLINICAL TRIAL: NCT03741491
Title: Birkebeiner II Study Investigating the Mechanisms of Atrial Fibrillation in Elderly Performing Endurance Training
Brief Title: Birkebeiner II Study
Status: Completed | Type: Observational
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Extrastiftelsen (Other)
Responsible Party: Principal Investigator, Marit Aarønæs, Head of outpatient clinic, Marit Aaronaes, MD, PhD, Diakonhjemmet Hospital
Other Study IDs: 2018/FO197570
Record Dates: First submitted 2018-11-02; First posted 2018-11-15 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples for DNA analysis and inflammation markers, Electronic ECG, Holter monitoring, Echocardiography
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Birkebeiner with AF: Persons already included in the Birkebeiner Aging Study (BIAS) (completed the Birkebeiner cross-country ski race in 2009/10 born 1945 and earlier) and BAF-study (completed the Birkebeiner cross-country ski race in 1999 and was born in 1960 and earlier) with AF.
- Birkebeiner without AF: Persons already included in the Birkebeiner Aging Study (BIAS) (completed the Birkebeiner cross-country ski race in 2009/10 born 1945 and earlier) and BAF-study (completed the Birkebeiner cross-country ski race in 1999 and was born in 1960 and earlier) without AF
- Control with AF: Persons included in HELMILO 2009 (Health and Environment Study in Oslo 2009), born 1960 and earlier with AF
- Control without AF: Persons included in HELMILO 2009 (Health and Environment Study in Oslo 2009), born 1960 and earlier without AF

SUMMARY:
Prolonged endurance exercise is associated with an elevated risk of atrial fibrillation (AF). The mechanisms governing this increased risk remains elusive. This study aim to detail the specific traits of elderly subjects with AF conducting endurance training by comparing elderly participators in the Birkebeiner cross country ski race(an indicator of prolonged endurance exercise practice) with and without AF to a not-so-trained control group.

DETAILED DESCRIPTION:
In recent years endurance sports with high intensity and participation in competition have been increasingly popular among middle aged and older people. The Birkebeiner studies are investigations of elderly non-professional athletes (65 years or older at enrollment in 2009/10) participating in the Birkebeiner cross-country ski race. It consists of Birkebeiner Aging Study, BIAS and the Birkebeiner Atrial Fibrillation, (BAF-study). The BAF-study investigated the association between prolonged endurance sport practice and the risk of AF by comparing the cohort of veteran cross-country skiers to a control population drawn from the Health and Environment Study in Oslo (HELMILO 2009).

The main findings of the Birkebeiner study so far have been that participation in the Birkebeiner cross-country ski race (an indicator of prolonged endurance exercise practice) is associated with an elevated risk of atrial fibrillation (AF) among men ≥ 65 years, and that this risk correlates with the cumulated amount of endurance-training. Similar findings were seen amongst female athletes. This increased risk of AF was shown independent of other known significant comorbidities (such as hypertension and diabetes), indicating that endurance-training at this level itself is an independent risk factor.

Regular physical exercise is an important factor when it comes to successful ageing. However, dose-relationship of physical exercise in a longer perspective is poorly studied. Atrial fibrillation is associated with increased risk of stroke, heart failure, dementia and death.

The mechanisms governing the increased risk of AF in elderly subjects undergoing endurance-training remains elusive. This study aim to detail the specific traits of elderly subjects with AF conducting endurance-training in comparison with trained and not-so-trained control groups. Thus, generating knowledge that can form the basis for better prevention and treatment of AF in this group.

ELIGIBILITY:
Inclusion Criteria:

* Already included in the Birkebeiner studies or "Health and environment study in Oslo" (HELMILO)
* Born 1960 and earlier

Exclusion Criteria:

* Born before 1935.
* Earlier heart valve surgery.
* MI (Mitral Insufficiency)≥ grade 3
* Ejection Fraction (EF) <35%

Ages: 58 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is drawn from earlier Birkebeiner studies and the Control Group from a Health population study in Oslo (HELMILO) matched by age and gender.
Sampling Method: Non-Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in atrial function and presence of atrial fibrillation in veteran endurance athletes | Cross sectional study. Measured at time for inclusion.
  Volume changes (ml) in the three phases of atrial function, measured by triplane echocardiography.
Changes in atrial function and presence of atrial fibrillation in veteran endurance athletes | Cross sectional study. Measured at time for inclusion.
  2D strain (%) in the three phases of atrial function, measured by triplane echocardiography.

SECONDARY OUTCOMES:
Changes in right ventricular volumes (ml) in veteran endurance athletes | Cross sectional study. Measured at time for inclusion.
  Measured by 2D echocardiography
Changes in p-wave (p-wave duration (msec), morphology and axis) in veteran endurance athletes | Cross sectional study. Measured at time for inclusion.
  Measured by ECG derived vector cardiograms.
Changes in R-R variability (msec) in veteran endurance athletes | Cross sectional study. Measured at time for inclusion.
  Measured by Holter ECG recordings
Presence of 171 genetic variants known to be associated with atrial fibrillation in veteran endurance athletes. | Cross sectional study. Measured at time for inclusion.
  Measured by genome-wide genotyping and next generation sequencing in the combination with Sanger sequencing.
Changes in biochemical markers associated with atrial fibrosis and inflammation in veteran endurance athletes. | Cross sectional study. Measured at time for inclusion.
  IL-1alfa, -1ra, -4,-6,-10, -17A, -17F, -21, -22, -23, -25, -31, -33, IFN-gamma TNF-alfa, IP-10, G-CSF, GM-CSF, MCP-1, MIP-1alfa, MIP-1beta, TIMP-1-4, MMP 1-3,7-10 and 12, measured by luminex multiplex technology
European Heart Rhythm Association (EHRA) score of atrial fibrillation related symptoms in veteran endurance athletes. | Cross sectional study. Measured at time for inclusion.
  Measured by European Heart Rhythm Association symptom score which is a classification of AF-related symptoms. The score ranges from I-no symptoms to IV-disabling symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Marit Aaronaes, MD,PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway